CLINICAL TRIAL: NCT05090839
Title: Expressing Personal Recollections in English or Spanish to Alleviate Traumatic Emotions (Exprésate)
Acronym: Exprésate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Roger McIntosh, Associate Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20190760; 5U54MD002266-15 (NIH)
Record Dates: First submitted 2021-10-12; First posted 2021-10-25 (Actual); Results first posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Post Traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Augmented trauma-writing intervention in Spanish (Experimental): Participants in this group will be required to write once weekly for 4 consecutive weeks. Participants will be instructed to write objectively about what they did the day prior and to avoid writing about their emotions or opinions in Spanish.
  Interventions: Behavioral: Weekly Emotional Disclosure (WED) Spanish
- Augmented trauma-writing intervention in English (Experimental): Participants in this group will be asked to write about their most traumatic or upsetting experiences for a total of 4 sessions (one session a week for 4 consecutive weeks) in English.
  Interventions: Behavioral: Weekly Emotional Disclosure (WED)
- Daily-event-writing control in English (Active Comparator): Participants in this group will be asked to conduct event writing condition in English and will be asked to write a description about what they did "yesterday from the time [they] got up until the time [they] went to bed" for 20 min continuously. They will be told to "avoid writing about [their] emotions or opinions" but to try to be as "accurate and objective as possible."
  Interventions: Behavioral: Weekly Emotional Disclosure (WED)
- Daily-event-writing control in Spanish (Active Comparator): Participants in this group will be asked to conduct event writing in condition in Spanish and will be asked to write a description about what they did "yesterday from the time [they] got up until the time [they] went to bed" for 20 min continuously. They will be told to "avoid writing about [their] emotions or opinions" but to try to be as "accurate and objective as possible."
  Interventions: Behavioral: Weekly Emotional Disclosure (WED) Spanish

INTERVENTIONS:
Behavioral: Weekly Emotional Disclosure (WED) — Online writing sessions, each lasting approximately 45 minutes, once a week, conducted virtually. Participants will be instructed to write about either a major traumatic life experience or what the participant did the previous day.
  Arms: Augmented trauma-writing intervention in English; Daily-event-writing control in English
Behavioral: Weekly Emotional Disclosure (WED) Spanish — Online writing sessions, each lasting approximately 45 minutes, once a week, conducted virtually. Participants will be instructed to write about either a major traumatic life experience or what the participant did the previous day in Spanish.
  Arms: Augmented trauma-writing intervention in Spanish; Daily-event-writing control in Spanish

SUMMARY:
The purpose of this study is to test if expressive writing about traumatic events has positive changes in women living with post-traumatic stress.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 21 years
2. Elevated PTSD symptoms as assessed by the Post-Traumatic Stress Disorder Checklist Scale-Version DSM 5 (PCL-5) using a cut-off of 34 or above
3. On a stable anti-retroviral therapy regimen for > 6 months as assessed with the Adult AIDS Clinical Trial Group structured interview
4. Spanish-English bilingual as measured by the Brief Acculturation Scale for Hispanics (cut-off of 3), Spanish speaker or English speaker
5. Participant is willing and able to sign Informed Consent Form (ICF)
6. self-report as Latina
7. HIV positive serostatus as determined by medical record within the last 12 months
8. Born female.

Exclusion Criteria:

1. Left-handedness or ambidextrous
2. Inability to tolerate the scanning procedures
3. Metal in body or prior history working with metal fragments
4. Any other contraindications for MRI examination (e.g., metallic implants such as pacemakers, surgical aneurysm clips, or known metal fragments embedded in the body)
5. currently pregnant or could be pregnant
6. Heavy alcohol intake (> 3 drinks) within 12 hours prior to participation in Functional Magnetic Resonance Imaging (fMRI)
7. Evidence from health history of neurological or systemic disorder which can cause cognitive impairment
8. Self-reported current diagnosis of psychiatric disorder or psychoactive substance abuse or dependence
9. Recent history (within two years) of myocardial infarction
10. Severe cardiovascular disease, or currently active cardiovascular disease (e.g., angina, cardiomyopathy)
11. Uncontrolled hypertension or hypotension
12. History of closed trauma with loss of consciousness
13. Space occupying lesions (e.g., mass lesions, tumors)
14. Central Nervous System (CNS) infection
15. CNS vasculitis
16. CNS demyelinating disease (e.g., multiple sclerosis)
17. Congenital CNS abnormality (e.g., cerebral palsy)
18. Seizure disorders
19. History of cerebrovascular disease (e.g., stroke, TIA's)

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-08-18 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-12-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger McIntosh, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited by flyers presented at community locations such as outpatient clinics, women's shelters, and at research centers located on the campus of the University of Miami.
Pre-assignment Details: Of the 40 participants enrolled, incomplete data collection resulted in 5 participants not being randomized and 6 were loss to follow-up prior to randomization. Thus, a total of 11 enrolled participants were not randomized.
Groups:
- Augmented Trauma-writing Intervention in Spanish: Participants in this group will be required to write once weekly for 4 consecutive weeks. Participants will be instructed to write objectively about what they did the day prior and to avoid writing about their emotions or opinions in Spanish.
  Weekly Emotional Disclosure (WED) Spanish Online writing sessions, each lasting approximately 45 minutes, once a week, conducted virtually. Participants will be instructed to write about either a major traumatic life experience or what the participant did the previous day. in Spanish.
- Augmented Trauma-writing Intervention in English: Participants in this group will be asked to write about their most traumatic or upsetting experiences for a total of 4 sessions (one session a week for 4 consecutive weeks) in English.
  Weekly Emotional Disclosure (WED) Online writing sessions, each lasting approximately 45 minutes, once a week, conducted virtually. Participants will be instructed to write about either a major traumatic life experience or what the participant did the previous day.
- Daily-event-writing Control in English: Participants in this group will be asked to conduct event writing condition in English and will be asked to write a description about what they did "yesterday from the time [they] got up until the time [they] went to bed" for 20 min continuously. They will be told to "avoid writing about [their] emotions or opinions" but to try to be as "accurate and objective as possible."
  Weekly Emotional Disclosure (WED) Online writing sessions, each lasting approximately 45 minutes, once a week, conducted virtually. Participants will be instructed to write about either a major traumatic life experience or what the participant did the previous day.
- Daily-event-writing Control in Spanish: Participants in this group will be asked to conduct event writing in condition in Spanish and will be asked to write a description about what they did "yesterday from the time [they] got up until the time [they] went to bed" for 20 min continuously. They will be told to "avoid writing about [their] emotions or opinions" but to try to be as "accurate and objective as possible."
  Weekly Emotional Disclosure (WED) Spanish Online writing sessions, each lasting approximately 45 minutes, once a week, conducted virtually. Participants will be instructed to write about either a major traumatic life experience or what the participant did the previous day in Spanish.
Period: Overall Study
Arm/Group | Augmented Trauma-writing Intervention in Spanish | Augmented Trauma-writing Intervention in English | Daily-event-writing Control in English | Daily-event-writing Control in Spanish
Started | 11 | 7 | 5 | 6
Completed | 9 | 4 | 4 | 5
Not Completed | 2 | 3 | 1 | 1
Not completed — Lost to Follow-up | 2 | 3 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Augmented Trauma-writing Intervention in Spanish: Participants in this group will be required to write once weekly for 4 consecutive weeks. Participants will be instructed to write objectively about what they did the day prior and to avoid writing about their emotions or opinions in Spanish.
  Weekly Emotional Disclosure (WED) Spanish Online writing sessions, each lasting approximately 45 minutes, once a week, conducted virtually. Participants will be instructed to write about either a major traumatic life experience or what the participant did the previous day in Spanish.
- Total: Total of all reporting groups
Arm/Group | Augmented Trauma-writing Intervention in Spanish | Augmented Trauma-writing Intervention in English | Daily-event-writing Control in English | Daily-event-writing Control in Spanish | Total
Number analyzed (Participants) | 11 | 7 | 5 | 6 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 7 | 5 | 6 | 29
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 5 | 6 | 29
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 6 | 5 | 6 | 28
  Not Hispanic or Latino | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1
  White | 11 | 6 | 5 | 6 | 28
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in PTSD Symptoms as Assessed by the Impact of Event Scale
Description: 22-item self-report instrument that corresponds to Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (DSM-IV) symptoms of PTSD over last 7 days on a scale from 0 (not at all) to 4 (extremely)
  The IES has a total score ranging from 0 to 88 with the higher score indicating greater PTSD symptoms. The IES was assessed before and after the intervention and the change in score (mean and SD) is reported as the outcome measure.
Time Frame: 6 weeks
Population: Data not analyzed from 19 participants that either did not complete a baseline or follow-up assessment of IES or who were lost to follow-up during the intervention.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Daily-event-writing Control in Spanish: Participants in this group will be asked to conduct event writing in condition in Spanish and will be asked to write a description about what they did "yesterday from the time [they] got up until the time [they] went to bed" for 20 min continuously. They will be told to "avoid writing about [their] emotions or opinions" but to try to be as "accurate and objective as possible."
  Weekly Emotional Disclosure (WED) Spanish Online writing sessions, each lasting approximately 45 minutes, once a week, conducted virtually. Participants will be instructed to write about either a major traumatic life experience or what the participant did the previous day.
Arm/Group | Augmented Trauma-writing Intervention in Spanish | Augmented Trauma-writing Intervention in English | Daily-event-writing Control in English | Daily-event-writing Control in Spanish
Number analyzed (Participants) | 11 | 7 | 6 | 5
score on a scale | -.383 (12.19) | 6.43 (4.27) | -3.18 (16.22) | -2.11 (9.59)
Statistical Analysis 1: Comparison: Augmented Trauma-writing Intervention in Spanish vs Augmented Trauma-writing Intervention in English; Test type: Equivalence — The 95% confidence interval is used to assess the difference between the means of the 2 x 2 (English vs. Spanish) and (Trauma vs. Non-trauma) writing groups; p < 0.05, ANOVA; variance explained by the IV. = .072, 95% CI 2-sided [.0000 to .234]

2. Primary Outcome: Changes in Verbal Learning as Assessed by Hopkins Verbal Learning Task
Description: Measures verbal learning and memory function based on the initial word learning list (0 no words recalled - 12 all words recalled).
Time Frame: baseline
Population: Data could not be collected at both timepoints due to time restraints and participant burden during. Hence, there was only one assessment of delayed recall performance on the HVLT.
Measure: Mean (Standard Deviation); unit: Total words recalled following delay.
Arm/Group | Augmented Trauma-writing Intervention in Spanish | Augmented Trauma-writing Intervention in English | Daily-event-writing Control in English | Daily-event-writing Control in Spanish
Number analyzed (Participants) | 7 | 3 | 2 | 5
Total words recalled following delay. | 10.43 (1.272) | 11.67 (.577) | 12 (.00) | 9.80 (1.92)

3. Secondary Outcome: Change in Functional Activity of the Default Mode Network (DMN).
Description: DMN is a large-scale network of interacting brain regions implicated in emotion and memory. Activity of the DMN hub indexed by Beta weight of activity within the ventral medial prefrontal cortex (VMPFC) was compared as a contrast between the visualizing trauma vs. visualizing stress conditions of the exposure. The VMPFC hub of the default mode network is a region integral to emotion regulation and is shown to be active during the use of cognitive-emotional regulation tasks (Andrewes and Jenkins, 2019). Hence, a randomization related increase in VMPFC activity while processing traumatic memories is associated with greater task engagement and cognitive-emotion regulation, which is a positive outcome.
Time Frame: 6 weeks
Population: Data not analyzed from 23 participants that either did not complete a baseline or follow-up fMRI assessment, or who's data could not be analyzed due to fMRI data not passing quality control (e.g., excessive motion, did not finish scan, signal distortion, etc.)
Measure: Mean (Standard Deviation); unit: Beta-weight reflecting change in BOLD
Arm/Group | Augmented Trauma-writing Intervention in Spanish | Augmented Trauma-writing Intervention in English | Daily-event-writing Control in English | Daily-event-writing Control in Spanish
Number analyzed (Participants) | 8 | 2 | 3 | 4
Beta-weight reflecting change in BOLD | .702 (.858) | -.716 (.906) | -.225 (.543) | -.118 (.762)
Statistical Analysis 1: Comparison: Augmented Trauma-writing Intervention in Spanish vs Augmented Trauma-writing Intervention in English; This is a comparison that is specific to the contrast of visualizing traumatic versus stressful events; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.05, ANOVA; Mean Difference (Final Values) = .358, 95% CI 2-sided [0 to .554]

4. Secondary Outcome: Change in Salivary Measures of Stress Reactivity.
Description: 200 uL of saliva will be used for immunosorbent assay of salivary alpha amylase (sAA) measured by picograms per milliliter
Time Frame: 6 weeks
Population: Data not analyzed from 29 participants that either did not complete a baseline or follow-up saliva collection or associated trauma recall tasks, were lost to follow-up during the intervention, had missing data from 1 of the three salivary time collection points, or samples not correctly recorded or collected.
Measure: Mean (Standard Deviation); unit: picograms per milliliter
Arm/Group | Augmented Trauma-writing Intervention in Spanish | Augmented Trauma-writing Intervention in English | Daily-event-writing Control in English | Daily-event-writing Control in Spanish
Number analyzed (Participants) | 1 | 3 | 3 | 4
picograms per milliliter | -871.9 (NA) — Only 1 participant in this cell. | -250.87 (11.9) | -622.3 (487.1) | -129.53 (267.15)
Statistical Analysis 1: Comparison: Augmented Trauma-writing Intervention in Spanish vs Augmented Trauma-writing Intervention in English; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.05, ANOVA; Mean Difference (Final Values) = .510, 95% CI 2-sided [.000 to .676]

ADVERSE EVENTS:
Time Frame: 2 years, 4 months
Description: Participants were provided with a measurement of SUDS (distress scale) before and after each session. This data and self-report was monitored for adverse effects.
Arm/Group | Augmented Trauma-writing Intervention in Spanish | Augmented Trauma-writing Intervention in English | Daily-event-writing Control in English | Daily-event-writing Control in Spanish
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/7 | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/7 | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 0/11 | 0/7 | 0/5 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-14): https://cdn.clinicaltrials.gov/large-docs/39/NCT05090839/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-17): https://cdn.clinicaltrials.gov/large-docs/39/NCT05090839/ICF_001.pdf